CLINICAL TRIAL: NCT01479361
Title: The Influence of Atazanavir-ritonavir and Efavirenz on Atovaquone Pharmacokinetics in HIV-infected Volunteers
Brief Title: Antiretroviral Drug Interaction Study in Volunteers With HIV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 120017; 12-CC-0017
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2016-06-01

CONDITIONS: HIV; PCP; Toxoplasmosis
Keywords: Atovaquone; Drug Interaction; Pharmacokinetics; Efavirenz; Atazanavir-Ritonavir; HIV
MeSH Terms: conditions — Toxoplasmosis | interventions — Atovaquone

INTERVENTIONS:
Drug: Atovaquone 750 mg twice daily
Drug: Atovaquone 1500 mg twice daily

SUMMARY:
Background:

- People who are infected with the human immunodeficiency virus (HIV) are at risk of getting certain diseases. Two of these diseases are a type of pneumonia known as PCP and a brain infection called toxoplasmosis. Most people with HIV take antiretroviral (ARV) drugs to treat HIV and lower the risk of infections. However, some ARV drugs may make other drugs used to treat PCP and toxoplasmosis less effective. Researchers want to test specific ARV drugs to see if they affect atovaquone, a drug used to treat PCP and toxoplasmosis.

Objectives:

- To see if ARV drugs atazanavir-ritonavir or efavirenz lower the blood levels of atovaquone.

Eligibility:

* Individuals between 18 and 70 years of age who have HIV.
* Participants must be taking efavirenz or atazanavir-ritonavir, or not taking any ARV drugs.

Design:

* Participants will be screened with a physical exam and medical history. They will also have blood and urine tests.
* This study has a screening visit and five study visits. Two of the study visits will last about 12 hours; the other three visits will last about 1 hour each.
* Participants will receive either a low dose or high dose of atovaquone to take for 14 days. They will record doses and any symptoms on a diary card at home.
* After 14 days, participants will have a 12-hour visit to provide blood samples. There will be a wash-out period with no doses for up to 6 weeks.
* After the wash-out period, participants will switch dose levels to either the high or low dose.
* After 14 days, participants will have a 12-hour visit to provide blood samples.

DETAILED DESCRIPTION:
The incidence of opportunistic infections such as Pneumocystis jirovecii pneumonia (PCP) and Toxoplasma gondii have substantially declined in patients with HIV infection due to potent combination antiretroviral (ARV) therapy and effective prophylaxis. The drug of choice for prophylaxis and treatment of PCP and toxoplasmosis is trimethoprim-sulfamethoxazole (TMP-SMX) and sulfadiazine, respectively. In patients who cannot tolerate these first line therapies, atovaquone is a common alternative. While generally considered safe and effective, a recent drug interaction study involving a single dose of combination tablet of atovaquone/proguanil (Malarone ) in HIV-infected patients showed that atovaquone plasma concentrations were significantly lowered (compared to healthy volunteers) by 75%, 74%, and 46% in patients taking the ARV medications efavirenz (EFV), lopinavir-ritonavir (LPV/r), and atazanavir-ritonavir (ATV/r), respectively. The mechanism of this drug interaction is unknown but is presumably due to induction of uridine diphosphate glucuronsosyltransferase (UGT) enzymes responsible for the metabolism of atovaquone. The magnitude of this interaction is such that it strongly suggests a clinically relevant drug interaction between atovaquone and the aforementioned ARVs. The purpose of this study is to determine whether HIV-infected subjects receiving ATV/r or EFV-containing ARV regimens, experience reductions in atovaquone exposure under steady state conditions compared to HIV-infected patients not receiving ARV therapy.

In this open-label study, 30 HIV-infected subjects will participate in 1 of 3 groups of 10 (Groups A, B, and C). Group A will consist of 10 subjects who are already receiving combination ARV therapy containing ATV/r; Group B will consist of 10 subjects already receiving combination ARV therapy containing EFV; and Group C will consist of 10 subjects who are not currently receiving ARV therapy. All subjects in Groups A, B, and C will be randomly assigned to either receive atovaquone 750 mg twice daily for 14 days (Phase 1) followed by a 2-6 week washout period, followed by atovaquone 1500 mg twice daily for 14 days (Phase 2), or vice versa. Pharmacokinetic (PK) sampling for atovaquone will occur on Day 14 of Phase 1 and 2.

Atovaquone PK parameters will be determined using non-compartmental methods with the WinNonlin professional computer program (version 5.2; Pharsight Corporation, Mountain View, CA). The following PK parameters will be compared among the groups: area under the concentration vs. time curve (AUC ?), maximum concentration (Cmax), apparent oral clearance (Cl/F), time to reach maximum concentration (Tmax), and half-life (T (Omega)). Data from this investigation will determine whether ATV/r and/or EFV alter the steady state PK of atovaquone in HIV-infected subjects. This information will assist clinicians in choosing appropriate alternative therapies for the treatment of PCP and toxoplasmosis in patients who are not candidates for first line therapies.

ELIGIBILITY:
* INCLUSION CRITERIA:

A subject will be considered eligible for this study only if all of the following criteria are met:

1. Between the ages of 18 and 70 years.
2. HIV-infected patients stabilized (greater than or equal to 90 days) on ARV regimens containing efavirenz 600 mg daily, or atazanavir/ritonavir 300/100 mg daily or HIV-infected patients not receiving ARV therapy.
3. CD4 cells greater than or equal to 350 cells/mm3 for HIV-infected patients not receiving ARV therapy.
4. CD4 cells >200 cells/mm3 for HIV-infected patients receiving ARV therapy.
5. Virologically suppressed patients receiving ARV therapy (<200 copies/mL on at least 2 consecutive occasions, within 6 months prior to enrollment).
6. Females of child bearing potential who are able and willing to prevent pregnancy by (a) practicing abstinence or (b) using effective methods of birth control, such as condoms, during the study period and for 1 month after study completion.
7. Subject agrees to storage of specimens for future research.

EXCLUSION CRITERIA:

A subject will be ineligible for this study if 1 or more of the following criteria are met:

1. Concomitant routine therapy with any prescription, over-the- counter, herbal, or holistic medications that are known or suspected to alter atovaquone including rifampin, rifabutin, and metoclopramide for 14 days prior to study participation.
2. Subjects receiving primary or secondary prophylaxis for PCP or toxoplasmosis.
3. ARV regimens containing both EFV and ATV/r.
4. Subjects receiving hormonal contraceptives within 90 days of Study Day 1.
5. Inability to obtain venous access for sample collection.
6. Laboratory and/or physical evidence of any active opportunistic infection.

   Diabetes mellitus requiring treatment with insulin, active tuberculosis, cardiac disease (uncontrolled hypertension and/or heart failure etc.), renal disease (chronic or acute renal failure or insufficiency resulting in baseline serum creatinine greater than 1.5 times upper limit of normal [ULN]), untreated/uncontrolled thyroid disease, untreated/uncontrolled psychiatric disease, active hepatitis (liver failure resulting in liver function tests greater than 3 times the ULN, ascites, or jaundice in the absence of ATV), or any other condition that may interfere with the interpretation of the study results or not be in the best interest of the subject in the opinion of the Investigator.
7. Positive pregnancy test or breastfeeding female.
8. The presence of persistent diarrhea or malabsorption that could interfere with the subject s ability to absorb drugs.
9. Drug or alcohol use that may impair safety or adherence.
10. History of intolerance or allergic reaction (rash; hives; swollen lips; difficulty breathing) to atovaquone.
11. Bleeding disorders (hemophilia, G.I., or intracranial bleeding).
12. Organ transplant recipient.
13. Documented ongoing problems with medication adherence.
14. High likelihood of switching ARV regimen within 12 weeks of the start of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-10-31; Primary Completion 2014-02-20 (Actual); Study Completion 2014-02-20 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to determine the steady state pharmacokinetics of 2 doses of atovaquone oral suspension in the presence of ATV/r, EFV, or no ARVs in HIV-infected patients.

SECONDARY OUTCOMES:
To compare our PK results with the recently reported interaction between a single dose of atovaquone+proguanil and ATV/r and EFV, and the comparator group which consists of HIV-infected subjects, as opposed to a comparator group of healthy subje...

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Kovacs, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Pifer LL, Hughes WT, Stagno S, Woods D. Pneumocystis carinii infection: evidence for high prevalence in normal and immunosuppressed children. Pediatrics. 1978 Jan;61(1):35-41. PMID 400818
- [Background] Hughes WT, Feldman S, Chaudhary SC, Ossi MJ, Cox F, Sanyal SK. Comparison of pentamidine isethionate and trimethoprim-sulfamethoxazole in the treatment of Pneumocystis carinii pneumonia. J Pediatr. 1978 Feb;92(2):285-91. doi: 10.1016/s0022-3476(78)80028-6. PMID 304478
- [Background] Winston DJ, Lau WK, Gale RP, Young LS. Trimethoprim-sulfamethoxazole for the treatment of Pneumocystis carinii pneumonia. Ann Intern Med. 1980 Jun;92(6):762-9. doi: 10.7326/0003-4819-92-6-762. PMID 6966901
- [Derived] Calderon MM, Penzak SR, Pau AK, Kumar P, McManus M, Alfaro RM, Kovacs JA. Efavirenz but Not Atazanavir/Ritonavir Significantly Reduces Atovaquone Concentrations in HIV-Infected Subjects. Clin Infect Dis. 2016 Apr 15;62(8):1036-1042. doi: 10.1093/cid/ciw028. Epub 2016 Jan 20. PMID 26797214